CLINICAL TRIAL: NCT06888414
Title: Evaluation of the Uterine Cavity by 3 D Ultrasonography in Perimenopausal Bleeding in Comparison With Hysteroscopy
Brief Title: Evaluation of the Uterine Cavity in Perimenopausal Women.
Status: Active, not recruiting | Type: Observational
Sponsor: Suez University (Other)
Responsible Party: Principal Investigator, Ahmed Sewidan, lecturer, Suez University
Other Study IDs: 1
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-03

CONDITIONS: Abnormal Uterine Bleeding, Unspecified
Keywords: 3D ultrasonography; Hysteroscopy
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Fifty perimenopausal women presenting with AUB were recruited from the outpatient clinic. Baseline data, including demographic, obstetric, and medical history, BMI, and laboratory investigations (CBC, renal and liver function tests, coagulation profile), were collected. All patients underwent transvaginal 3D ultrasonography and hysteroscopy.
  Interventions: Diagnostic Test: transvaginal ultrasound

INTERVENTIONS:
Diagnostic Test: transvaginal ultrasound — Fifty perimenopausal women presenting with AUB were recruited from the outpatient clinic. Baseline data, including demographic, obstetric, and medical history, BMI, and laboratory investigations (CBC, renal and liver function tests, coagulation profile), were collected. All patients underwent transvaginal 3D ultrasonography and hysteroscopy.

SUMMARY:
Abnormal uterine bleeding (AUB) in perimenopausal women is a common yet poorly defined condition requiring accurate diagnosis. Hysteroscopy is the gold standard for evaluating intrauterine abnormalities, but 3D ultrasonography (3D US) has emerged as a non-invasive alternative.

DETAILED DESCRIPTION:
Change in menstrual blood volume is a common manifestation of perimenopause, often indicative of underlying gynecological conditions. The etiology of perimenopausal bleeding is multifactorial and may include hormonal imbalances, endometrial polyps, malignancies, adenomyosis, vascular malformations, and systemic medical conditions.

The evaluation of uterine pathology can be achieved through both invasive and non-invasive diagnostic modalities. Ideally, non-invasive techniques are preferred due to their safety, cost-effectiveness, and ease of use. Ultrasonography is considered a reliable, non-invasive imaging tool for assessing uterine abnormalities and is often employed as a preliminary diagnostic step before invasive procedures such as hysteroscopy.

Among invasive techniques, hysteroscopy remains the gold standard for direct visualization of the uterine cavity. This method enables precise assessment of intrauterine pathology, facilitating accurate diagnosis and treatment planning. Compared to other imaging modalities, such as hysterosalpingography, hysteroscopy provides superior diagnostic accuracy and therapeutic potential.

Non-invasive diagnostic approaches, including transabdominal ultrasound (TAS) and two-dimensional transvaginal sonography (2D-TVS), are widely utilized in evaluating abnormal uterine bleeding (AUB). These modalities help detect uterine lesions such as fibroids, polyps, and focal abnormalities while also assessing adnexal pathology. Three-dimensional ultrasonography (3D-US) further enhances diagnostic capabilities by allowing multiplanar reconstruction from volumetric data, improving visualization of the endometrial cavity and providing a more detailed assessment of uterine morphology.

Three-dimensional transvaginal sonography (3D-TVS) is a cost-effective, non-invasive, and highly efficient method for indirectly visualizing the endometrial cavity. Given its accessibility and diagnostic accuracy, it is recommended as a first-line imaging modality for evaluating uterine lesions in reproductive-aged women presenting with abnormal uterine bleeding.

Despite advancements in diagnostic imaging, there remains a gap in knowledge regarding the optimal use of 3D transvaginal ultrasonography (3D-TVS) as a standalone tool for diagnosing intrauterine pathology. While hysteroscopy is the gold standard, further research is needed to refine the sensitivity and specificity of 3D-TVS in differentiating benign from malignant lesions, reducing the need for unnecessary invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 -55 years.
* Patients complaining of abnormal uterine bleeding not receiving hormonal treatment for the last three months or intrauterine device as it affects the endometrial thickness by ultrasound and the accuracy of the pathology.
* Free from chronic medical diseases: renal, liver, chest and heart diseases.

Exclusion Criteria:

* Age less than 40 and more than 55 years.
* Patients received hormonal treatment.
* Patients with chronic diseases or have coagulopathy.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Perimenopausal patients with presented to the outpatient clinic with abnormal uterine bleeding
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of 3 D ultrasound in diagnosis of uterine causes perimenopausal bleeding versus hysteroscopy | 3 months
  Sensitivity and specificity of transvaginal ultrasound versus hysteroscopy in diagnosis perimenopausal bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Suez university, Suez, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lalchandani S, Phillips K. Evaluation of endometrial cavity-investigation options. Reviews in Gynaecological Practice. 2003 Sep 1;3(3):165-70. https://doi.org/10.1016/S1471-7697(03)00065-0
- [Result] Clinico histopathological evaluation of abnormal uterine bleeding in women of reproductive and perimenopausal age group